CLINICAL TRIAL: NCT03440008
Title: Improving the Detection, Classification and Treatment of Misaligned Arthritic Ankles
Acronym: IDCT
Status: Terminated | Type: Observational
Why Stopped: As a consequence of the COVID-19 pandemic, this study was first paused then ended as the PI moved to a different service line over the course of the VHA's COIVD-19 response.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F2318-W
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Ankle Osteoarthritis
MeSH Terms: interventions — Foot Orthoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: None Retained — No biospecimens will be collected for this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Able-bodied, age matched subjects with no foot and ankle pathology
  Interventions: Other: Dynamic 3D bone motion capture
- OA: Subjects with ankle OA, with all classifications of ankle misalignment (varus, neutral, valgus)
  Interventions: Other: Dynamic 3D bone motion capture; Device: wedged insole

INTERVENTIONS:
Other: Dynamic 3D bone motion capture — Two x-ray systems will image the subjects ankle while they walk, allowing us to calculate ankle joint angle and alignment
  Other Names: Biplane fluoroscopy
Device: wedged insole — medial or lateral wedge (appropriate for varus or valgus misalignment) will be applied during 1 data collection session to evaluate effect of wedging on misalignment
  Other Names: orthotic/insole
  Groups: OA

SUMMARY:
The Veteran population is prone to foot and ankle maladies from common injuries such as sprains, and diseases such as ankle osteoarthritis (cartilage damage). More specific to Veterans are prior service injuries of the foot and ankle, which historically account for nearly a quarter of injuries received. These injuries include bone fractures and ligament damage. Some of these injuries may lead to poor ankle joint alignment, which over time could lead to osteoarthritis due to abnormal wear on a day to day basis. The goal of this proposal is to use a novel technology - biplane fluoroscopy, to study the movement of ankles which are misaligned in subjects with ankle osteoarthritis. This proposal will also benefit current diagnostic methods with additional information. Last, this proposal will test the effectiveness of a conservative treatment (modified shoe insoles) to correct or reduce the misalignment in ankles. This proposal will create evidence about: the nature of ankle osteoarthritis, the accuracy of diagnosing alignment, and conservative treatment for patients with ankle OA.

DETAILED DESCRIPTION:
Ankle osteoarthritis (OA) is a debilitating and mobility limiting condition. It can commonly stem from the result of a traumatic injury - such trauma has a high prevalence in military service. If cartilage is not severely damaged in that trauma, the stability and alignment of the joint may be. Over time, an unstable or misaligned ankle joint can experience abnormal rates of cartilage wear and tear due to aberrant kinematics. While OA may take decades to develop, the resulting arthritic state from this trauma will ultimately require ankle replacement or fusion, consequences with a tremendous financial burden and quality of life impact.

With regards to alignment, particularly in the coronal plane, current clinical diagnosis relies on static X-ray of the ankle joint. Static images may not indicate dynamic misalignment during gait. Further, the effect of wedged insoles, a potential conservative treatment, on the restoration of ankle function is undocumented.

This proposal aims to use biplane fluoroscopy, an X-ray based dynamic imaging approach, to measure ankle kinematics in OA subjects (with varus, neutral and valgus ankle alignment) and controls. With this method, tibio-talar kinematics during gait can be measured. Furthermore, subjects classified as neutral from their static radiograph, but that exhibit ankle varus or valgus alignment during gait, will be identified. Improving the accuracy of a diagnostic outcome provides a patient group with additional avenues for treatment. The investigators will investigate correlations between the investigators' 3D kinematics and clinical 2D imaging - to the benefit of clinical diagnostics. The investigators will also be able to measure the effect of wedged insoles on the restoration of ankle function. With this in mind, the following aims and methodology are proposed.

Specific Aim 1: To investigate ankle kinematics in controls and subjects with OA. In support of Specific Aim 1, 90 ankle OA subjects will be recruited (30 each of varus, neutral or valgus aligned ankles). The investigators will also recruit 20 control subjects. Subjects will receive CT scans of their feet to quantify bone geometry (a step necessary for biplane fluoroscopy). Subjects will then be imaged in the biplane system during gait trials and while wearing neutral study shoes. This will yield tibio-talar kinematics during gait for these populations. Specific Aim 2: To identify dynamically misaligned ankles in OA subjects who are currently classified as neutrally aligned using static analysis. The investigators will compare the static X-ray and the gait kinematics of OA subjects, particularly those with clinically determined neutral alignment. The investigators will determine what proportion of neutral OA subjects actually exhibit misalignment during gait and are thus improperly categorized. The investigators will also re-create 2D clinical X-ray views from the investigators' 3D data in an attempt to translate the investigators' improvement (with 3D fluoroscopy) to more accurately classify alignment to clinical 2D diagnostics. Specific Aim 3: To evaluate the potential of lateral or medial wedging to restore alignment in misaligned ankle OA subjects. OA subjects will be imaged wearing shoes with wedged insoles which correspond to their type of misalignment. Neutral OA subjects, who demonstrate misalignment during gait, will be recalled for a wedged insole session. This yields conservative treatment kinematics.

This study will generate baseline data describing the kinematics of control and ankle OA subjects. This data is not currently available in the literature, and represents a novel contribution to the field. Second, this proposal determines how accurate current 2D X-ray methods are at detecting dynamic misalignment. This information can inform clinicians about the accuracy of their diagnostic tools, and may lead to improvements. Third, this proposal will generate data to evaluate the utility of wedged insoles for the conservative management of ankle misalignment. In Summary, this study has immediate impact potential on the diagnosis and treatment of ankle OA. Last, there are numerous additional avenues of classification, diagnostic, and preventative research for the benefit of the Veterans which will stem from this Career Development Award.

"As a consequence of the COVID-19 pandemic, and after consultation with the appropriate research oversight, regulatory and monitoring entities, screening and enrollment has been placed on temporary administrative hold as of 03/16/2020."

ELIGIBILITY:
Inclusion Criteria:

* Be ambulatory (able to walk at least 15 m, and tolerate ~1 hour of standing and walking with rest periods)

Exclusion Criteria:

* Recent (<1 year) surgical, neurological, metabolic or lower limb musculoskeletal problem that might impair the ambulation measures in the study

  * Such as severe knee or hip osteoarthritis
* Diagnosed with diabetes, peripheral neuropathy, or peripheral vascular disease
* For OA subjects, a radiographic discontinuity of the cartilage of the tibial plafond or talar dome
* Also for OA subjects, rapid onset of OA (<3 years) following ankle fracture
* Diagnosis of severe ankle instability or deformity such as pes planus
* Inadequate cognitive or language function to consent or to participate

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Controls and those with ankle osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2023-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Iaquinto, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a combination of clinician introduction to the study, and posted recruitment materials in 2 hospital systems (VA and academic). The study was open for recruitment in 2016 but due to a laboratory move and hardware update, the first participant was not enrolled until February 2019. The last participant was enrolled in March 2020, three days before a local hold on in-person research was enacted due to the COVID-19 pandemic.
Pre-assignment Details: Of 33 enrolled participants, 32 proceeded into either control or OA cohorts, one participant withdrew.
Groups:
- OA (Osteoarthritis): Subjects with ankle OA, with all classifications of ankle misalignment (varus, neutral, valgus)
  Dynamic 3D bone motion capture: Two x-ray systems will image the subjects ankle while they walk, allowing us to calculate ankle joint angle and alignment
  wedged insole: medial or lateral wedge (appropriate for varus or valgus misalignment) will be applied during 1 data collection session to evaluate effect of wedging on misalignment
Period: Overall Study
Arm/Group | Control | OA (Osteoarthritis)
Started | 26 | 7
Completed | 0 | 0
Not Completed | 26 | 7
Not completed — Cessation of research visits due to COVID-19, PI was transferred to a crisis-response department | 25 | 7
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | OA (Osteoarthritis) | Total
Number analyzed (Participants) | 25 | 7 | 32
Age, Continuous [Mean (Full Range); unit: Years] | 59.0 [41 to 78] | 55.4 [38 to 68] | 58.2 [38 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 0 | 12
  Male | 13 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 23 | 5 | 28
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 0 | 6
  White | 17 | 4 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 7 | 32
Varus/Neutral/Valgus Alignment [Count of Participants; unit: Participants]
  Varus Misaligned | 0 | 0 | 0
  Neutral Alignment | 0 | 0 | 0
  Valgus Misaligned | 0 | 0 | 0
  Unknown Alignment | 25 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Tibio-talar Kinematics During Gait
Description: The 3D movement between the tibia and talus bones will be assessed using biplane fluoroscopy, for OA and control subjects during shod gait.
Time Frame: 4 hour session
Population: Differences in 6 degree-of-freedom motion between the tibia and talus during shod gait (contact phase), between Controls and OA participants. Note that this study was terminated before this data was collected, thus no analysis is available.
Arm/Group | Control | OA (Osteoarthritis)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Static Ankle Alignment Sensitivity
Description: The sensitivity to correctly diagnose dynamic misalignment by using static x-ray images, will be determined for the OA population.
Time Frame: 4 hour session
Population: For OA participants, differences between their static alignment classification, and their dynamically measured varus / neutral / valgus status. Note that this study was terminated before this data was collected, thus no analysis is available.
Arm/Group | Control | OA (Osteoarthritis)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Decrease in Misalignment During Gait Using Wedged Insoles
Description: The effect that wedged insoles have on varus / valgus misalignment will be assessed using dynamic 3D x-ray
Time Frame: 4 hour session
Population: Measure of changes in coronal plane tibio-talar motion in OA population with and without wedged insoles. Note that this study was terminated before this data was collected, thus no analysis is available.
Arm/Group | Control | OA (Osteoarthritis)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No participants performed any study visits (e.g. for Primary Outcome 1-3), therefore there were no periods of time over which AE, SAE, or UAPs could be collected.
Description: "0" Total Number of Participants at Risk (e.g., serious and other [non-serious] adverse events were not collected or assessed as part of the study).
Arm/Group | Control | OA (Osteoarthritis)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03440008/Prot_SAP_000.pdf